CLINICAL TRIAL: NCT06617871
Title: A Prospective, Randomized, Single-blinded Clinical Trial Comparing Mechanical Alignment Vs Kalipered Kinematic Alignment Total Knee Arthroplasty Using Medacta Spherika
Brief Title: Mechanical Alignment Vs Kalipered Kinematic Alignment Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Medacta International SA (Industry)
Responsible Party: Principal Investigator, Adam Edelstein, Assistant Professor of Orthopaedic Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00219231
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Knee Osteoarthritis; Knee Arthropathy
Keywords: randomized trial; knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Methods

STUDY DESIGN:
Intervention Model Description: 1:1
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mechanical Alignment (MA) (Active Comparator): Primary TKA with the Medacta SpheriKA, utilizing either MA methodology.
  Interventions: Procedure: Mechanical Alignment (MA)
- Kinematic Alignment (KA) (Active Comparator): Primary TKA with the Medacta SpheriKA, utilizing either KA methodology.
  Interventions: Procedure: Kinematic Alignment (KA) Interventions:

INTERVENTIONS:
Procedure: Mechanical Alignment (MA) — Primary TKA with the Medacta SpheriKA, utilizing either MA methodology.
  Arms: Mechanical Alignment (MA)
Procedure: Kinematic Alignment (KA) Interventions: — Primary TKA with the Medacta SpheriKA, utilizing either KA methodology.
  Arms: Kinematic Alignment (KA)

SUMMARY:
Knee replacement surgery can be performed in one of two ways. Traditionally the goal was for the new joint to be in a neutral position with respect to the femur (thigh bone). This is called Mechanical Alignment (MA). The neutral position is different than the human knee's natural position, so MA often requires the surgeon to make additional cuts to the ligaments and other soft tissue around the knee. More recently surgeons have started to place the new joint in a position that more closely replicates the natural alignment of the human knee. This is called Kinemetic Alignment (KA). KA can be done without additional soft tissue dissection but the procedure requires a higher level of precision that can be difficult to achieve in every case.

Some studies have found no difference in outcomes between MA and KA, whereas others have found KA to be superior. But these were small studies or studies that did not consider patient-rated outcomes.

DETAILED DESCRIPTION:
Up to 20% of patients that report dissatisfaction and chronic pain following Total knee arthroplasty (TKA). Prior research has identified patient demographic, comorbidity, and expectations as factors that are associated with dissatisfaction. Emerging literature has also suggested that surgical factors including component alignment, soft tissue balance, and kinematics may play a role in patient satisfaction, and that modifications to alignment may result in better function than performing soft tissue releases. Personalized alignment strategies have been proposed that aim to more closely recreate native knee morphology and kinematics. Kinematic alignment (KA) describes a technique that aims to restore the pre-arthritic joint surfaces and alignment of the femur and tibia by removing the bone and cartilage thickness that will be replaced by the implant, taking into account cartilage wear. KA can therefore be conceptualized as a resurfacing procedure, wherein native joint surfaces are replaced by prosthetic surfaces but the position and alignment of the joint surfaces are not changed. This contrasts with mechanical alignment (MA), in which implants are positioned perpendicular to the mechanical axes of the femur and tibia in a manner independent of the pre-arthritic joint surfaces, and soft tissue releases are performed to bring limb alignment into mechanical neutral.

There have been prior randomized trials comparing kinematic and mechanical alignment, and these have had mixed results regarding the superiority of one approach over the other. The majority of these trials did not use the same operative modality for both groups (manual vs computer-assisted techniques) or did not include relevant patient reported outcomes (PROs). There is a need for a prospective, randomized trial comparing outcomes following kinematic vs mechanical alignment TKA, with the same operative modality used in both groups with inclusion of relevant PROs.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing primary TKA with a medially-stabilized SpheriKA knee system
* Able to read and understand consent form and PRO instruments and willing to return for follow up visits

Exclusion Criteria:

* Varus or Valgus malalignment >15 degrees to mechanical axis
* Flexion contracture >15 degrees or flexion <90 degrees
* BMI >40
* Revision TKA or other prior knee surgery other than arthroscopy or arthroscopic-assisted ligament reconstruction
* Diagnosis or history of any of the following

  * inflammatory arthritis
  * infection in study knee
  * chronic pain
  * chronic opioid use
  * metabolic musculoskeletal disorder other than osteopenia/osteoporosis
* Patients receiving workers' compensation for study condition
* Patients who cannot complete questionnaires in English
* Patients with comorbidities preventing surgery
* Patients who are not able to provide informed consent

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
6-week Knee Injury and Osteoarthritis - Joint Replacement Score (KOOS-JR) | 6 weeks postoperative
  The Knee Injury and Osteoarthritis Score - Joint Replacement (KOOS-JR) score

SECONDARY OUTCOMES:
Forgotten Joint Score (FJS) | 1 year postoperative
  Forgotten Joint Score (FJS) questionnaire score

CONTACTS AND LOCATIONS:
Overall Officials: Adam Edelstein, MD, Principal Investigator — Assistant Professor of Orthopaedic Surgery
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregate data will be shared via ClinicalTrials.gov
Supporting Information: Study Protocol, ICF
Time Frame: Supporting information will be available after all manuscripts have been published.
Access Criteria: Contact study PI